CLINICAL TRIAL: NCT03649256
Title: Deficient Lower Segment Cesarean Section Scar, Does the Type of Suture Matter?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, David Peleg, Staff physician, Ziv Hospital
Other Study IDs: ZIV-0085-18
Record Dates: First submitted 2018-08-21; First posted 2018-08-28 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: 2 Arms, Conventional Suture, Barbed Suture
Keywords: conventional suture, barbed suture, niche, scar, cesarean section
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Conventional suture: closure of uterine incision with conventional suture (Vicryl, Ethicon)
  Interventions: Diagnostic Test: Thickness of lower uterine segment scar
- Barbed suture: closure of uterine incision with barbed suture (Stratafix, Ethicon)
  Interventions: Diagnostic Test: Thickness of lower uterine segment scar

INTERVENTIONS:
Diagnostic Test: Thickness of lower uterine segment scar — Ultrasound measurement of thickness of the uterine scar at 3 and 6 months

SUMMARY:
In recent years there has been a significant increase in cesarean sections. This is not without complication in subsequent pregnancies such as placenta previa, placenta accrete, scar pregnancy, dehiscence or uterine rupture. Uterine rupture during trial of labor after cesarean section is an uncommon but potentially catastrophic, life threatening event. It is thus of importance if the investigators were able to predict the risk of uterine rupture. Imaging studies including ultrasound, hysterography and sonohysterography have been used to evaluate the scar from a prior cesarean before pregnancy, there is no consensus as to which of them is the preferred method but it is known that cesarean section scars can be detected reliably by ultrasound imaging. Previous studies have shown that sonographic lower uterine segment thickness is a strong predictor for uterine scar defect and could represent a high risk of uterine rupture during a trial of labor in women with prior cesarean section. There is a likely association between large defects in the scar after cesarean delivery detected by transvaginal ultrasonography in non pregnant women and uterine rupture or dehiscence in subsequent pregnancy.

The knotless barbed suture was FDA approved in 2004. Knotless barbed sutures are monofilament sutures with barbs cut into them. These sutures self-anchor, maintaining tissue approximation without the need for surgical knots.

The objective of this study is to determine whether there is a difference in the lower uterine segment thickness between uterine scars sutured with two types of sutures, to determine whether there is a difference in the size of the scar defects.

Methods: Two hundred and two women will undergo transvaginal ultrasound examination 3 and 6 months after delivery: 101 women will have undergone cesarean section in which the Vicryl suture was used, 101 women will have undergone cesarean section in which the KBS suture was used. The ultrasound examiner will be blinded to the use of the suture. The investigators will measure the myometrial thickness 3 months and 6 months after the delivery and compare the results between the 2 groups.

The assumption is that the findings of the study will be useful in counseling concerning Trial of Labor after Cesarean (TOLAC). To the best of the investigators' knowledge, there are no published data on the risk of uterine rupture predicted based on the myometrial thickness measured in the non-pregnant patient when the knotless barbed suture was used in the cesarean section. Previous studies have examined the applicability of low uterine segment measurement in the third trimester in the prediction of a uterine defect during trial of labor

ELIGIBILITY:
Inclusion Criteria:

* Post Cesarean section

Exclusion Criteria:

* Non low- transverse incision, after myomectomy, pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: status post cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 202 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Uterine Thickness | 6 months
  uterine myometrial thickness as measured by ultrasound

SECONDARY OUTCOMES:
Uterine Thickness | 3 months
  uterine myometrial thickness as measured by ultrasound

IPD SHARING:
Plan to Share IPD: No